CLINICAL TRIAL: NCT07228091
Title: Surgical Procedure Efficiency Evaluation stuDy (SPEED): Combination Phaco-Vitrectomy Surgeries With UNITY VCS vs. Constellation in a Real-World Operating Room Setting
Brief Title: Surgical Procedure Efficiency Evaluation stuDy
Status: Not yet recruiting | Type: Observational
Sponsor: Alcon Research (Industry)
Collaborators: Manchester Royal Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CTV678-H003
Record Dates: First submitted 2025-11-12; First posted 2025-11-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Cataract; Vitreous Hemorrhage; Retinal Detachment; Macular Pucker; Macular Holes
Keywords: anterior segment ophthalmic surgery; posterior segment ophthalmic surgery
MeSH Terms: conditions — Cataract; Vitreous Hemorrhage; Retinal Detachment; Epiretinal Membrane; Retinal Perforations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- UNITY VCS: Subjects will undergo routine scheduled combined anterior-posterior segments surgery (phacovitrectomy)
  Interventions: Device: UNITY VCS
- CONSTELLATION: Subjects will undergo routine scheduled combined anterior-posterior segments surgery (phacovitrectomy)
  Interventions: Device: CONSTELLATION

INTERVENTIONS:
Device: UNITY VCS — UNITY® VCS is a CE-marked, FDA-approved ophthalmic microsurgical system that is indicated for both anterior segment (i.e., phacoemulsification and removal of cataracts) and posterior segment (i.e., vitreoretinal) ophthalmic surgery. The focus of this study will be on combined anterior-posterior segments surgery (phacovitrectomy).
  Other Names: UNITY® Vitreoretinal Cataract System (VCS)
  Groups: UNITY VCS
Device: CONSTELLATION — CONSTELLATION is a CE-marked, FDA-approved ophthalmic microsurgical system that is indicated for both anterior segment (i.e., phacoemulsification and removal of cataracts) and posterior segment (i.e., vitreoretinal) ophthalmic surgery. The focus of this study will be on combined anterior-posterior segments surgery (phacovitrectomy).
  Other Names: CONSTELLATION® Vision System
  Groups: CONSTELLATION

SUMMARY:
The purpose of this real-world evidence study is to compare surgical procedure times for UNITY® VCS and CONSTELLATION® Vision System.

DETAILED DESCRIPTION:
Eligible subjects will undergo routine scheduled combined anterior-posterior segments surgery (phacovitrectomy). This single visit, time-and-motion study will be conducted in the United Kingdom. This study will be conducted by Alcon Vision LLC.

ELIGIBILITY:
Key Inclusion Criteria:

* Able to understand and sign an informed consent form (ICF) that has been approved by an ethics committee.
* Planned combined phacovitrectomy procedure at one of the selected surgical sites.
* Planned combined phacovitrectomy procedure with 25-gauge (G) vitrectomy tools.

Key Exclusion Criteria:

* Unplanned/emergency phacovitrectomy.
* Pregnant.
* Past history of phacovitrectomy. cataract, vitrectomy in the planned operative eye.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the clinical practice of the participating Investigator.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of surgeons replying "efficient" or "very efficient" to the question, "How would you rate overall OR (operating room) efficiency of the console for the combined phaco-vitrectomy surgery (including set-up/tear-down)? | Up to Day 1 post completion of the surgery
  Responses will be collected on a 5-point scale where 1=Very Inefficient, 2=Inefficient, 3=Neutral, 4=Efficient, and 5=Very Efficient.

CONTACTS AND LOCATIONS:
Overall Officials: Manager, Health Economics/Outcomes Research, Study Director — Alcon Research, LLC
Locations (2):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States
- Manchester Royal Eye Hospital, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No